CLINICAL TRIAL: NCT01715753
Title: Does Enhanced Protein Intake Preserve Function and Lean Muscle Mass During Weight Reduction in Frail, Obese Older Adults?
Brief Title: Measuring Eating, Activity and Strength: Understanding the Response -Using Protein
Acronym: MEASUR-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00037110; 3834193 (Other Grant/Funding Number: National Cattlemen's Beef Association)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-03

CONDITIONS: Weight Loss
Keywords: Function; Muscle mass
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight Loss Control (Active Comparator): Diet counseling and group education lessons. Subjects follow a calorie-reduction diet for a weight loss of ≥10%.
  Interventions: Behavioral: Diet counseling and group education lessons
- Weight Loss-High Protein (Experimental): Protein supplementation. Subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of protein, including substantial amounts of supplemental protein provided as lean beef. Intakes of > 30g of high quality protein will be achieved three times a day by subjects in this group, with all or predominantly all from animal source and 60-70% of animal protein from beef.
  Interventions: Dietary Supplement: Protein supplementation

INTERVENTIONS:
Dietary Supplement: Protein supplementation — > 30g of high quality protein will be achieved three times a day by subjects in this group, with all or predominantly all from animal source and 60-70% of animal protein from beef.
  Arms: Weight Loss-High Protein
Behavioral: Diet counseling and group education lessons — Individual and group diet counseling to achieve a >10% weight loss
  Arms: Weight Loss Control

SUMMARY:
The purpose of the trial is to assess the effects of weight loss on functional status and lean muscle mass in frail, obese older adults (>/= 60) who participate in a 6 month weight reduction intervention. Participants will be randomized into one of two study arms: Weight Loss Control: (n = 25) subjects follow a calorie-reduction diet for a weight loss of ≥10%; or Weight Loss-High Protein: (n = 50) subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of high quality protein at each meal. Intakes of > 30g of high quality protein will be achieved three times a day by subjects in this group, predominantly all from animal sources and 60-70% of animal protein from beef. Subject criteria will include obese (>30 kg/m2) older adults (>60 yrs.) with mild to moderate functional impairment (by Short Physical Performance Battery; SPPB score >/= 4)

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ yrs.
* BMI of >30 kg/m2
* Body weight <495 lbs.
* Normal blood chemistries
* Normal renal function
* Primary care physician acknowledgement
* Non-Vegetarian
* Mild to moderate movement impairment

Exclusion Criteria:

* Body weight >495 pounds.
* Current smoker.
* Presence of unstable, acutely symptomatic, or life-limiting illness.
* Positive screen for dementia using Mini-Cog evaluation tool.
* Neurological conditions causing functional or cognitive impairments.
* History of significant weight instability (defined as > 10 pounds weight gain or loss over 6 months prior to study participation).
* Unwillingness or inability to be randomized to any one of two intervention groups, submit to all study testing or continuously participate in a randomly assigned lifestyle intervention program for six months.
* Inability to walk independently.
* Bilateral hip replacements.
* Unable to give consent.
* Unable to complete written recording forms including journals of eating and exercise behaviors.
* Current use of the following medications: monoamine oxidase inhibitors, prescription weight loss medications.
* Primary Care Physician advises against participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) | Baseline to 3 to 6 months
  short physical performance battery
Change in lean body mass | Baseline to 3 and 6 months
  Bodpod

OTHER OUTCOMES:
Change in baseline lipids (classes, subclasses, participle size and number) at 6 months | Baseline to 6 months
  Concentrations for lipoprotein classes (VLDL, LDL and HDL particle numbers) and subclasses (small, medium and large) were calculated using the LP3 deconvolution algorithm. Mean VLDL, LDL and HDL particle sizes were weighted averages derived from the sum of the diameter of each subclass multiplied by its relative mass percentage.
Changes in baseline GlycA at 6 months | Baseline to 6 months
  NMR-measured systemic inflammatory factor and a biomarker of CVD risk
Change in baseline trimethylamine-N-oxide (TMAO) at 6 months | Baseline to 6 months
  TMAO is a metabolite produced from trimethylamine (TMA) containing nutrients. Nuclear magnetic resonance (NMR) spectroscopy assay was used for quantification of TMAO concentrations.
Change in baseline betaine at 6 months | Baseline to 6 months
  Betaine was measured by 1H-nuclear magnetic resonance (NMR) spectroscopy using a Vantera® NMR Clinical Analyzer (LabCorp, Raleigh, NC).
Change in baseline branched chain amino acids (BCAA) at 6 months | Baseline to 6 months
  NMR MetaboProfile analysis, which reports concentrations of several metabolites [ the branched chain amino acids (BCAA) valine, leucine, and isoleucine] was performed using the recently developed LP3 deconvolution algorithm.
Change in baseline Lipoprotein Insulin Resistance Index (LP-IR) scores at 6 months | Baseline to 6 months
  LP-IR is a composite metabolomic biomarker that captures the multidimensional effects of insulin resistance on the lipoprotein metabolic chain. It is measured by nuclear magnetic resonance spectroscopy as a weighted score of VLDL, LDL and HDL particle sizes, and their subsets concentrations.
Change in baseline GFR at 6 months | Baseline to 6 months
  Estimated GFR, which measures renal filtering capacity, is a calculated value based on age, sex, race, and serum creatinine using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
Change in baseline fasting glucose at 6 months | Baseline to 6 months
  Level of glucose in the blood after fasting for at least 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Connie W Bales, PhD, RD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Porter Starr KN, Orenduff M, McDonald SR, Mulder H, Sloane R, Pieper CF, Bales CW. Influence of Weight Reduction and Enhanced Protein Intake on Biomarkers of Inflammation in Older Adults with Obesity. J Nutr Gerontol Geriatr. 2019 Jan-Mar;38(1):33-49. doi: 10.1080/21551197.2018.1564200. Epub 2019 Feb 27. PMID 30810500
- [Derived] Payne ME, Porter Starr KN, Orenduff M, Mulder HS, McDonald SR, Spira AP, Pieper CF, Bales CW. Quality of Life and Mental Health in Older Adults with Obesity and Frailty: Associations with a Weight Loss Intervention. J Nutr Health Aging. 2018;22(10):1259-1265. doi: 10.1007/s12603-018-1127-0. PMID 30498835
- [Derived] Porter Starr KN, Pieper CF, Orenduff MC, McDonald SR, McClure LB, Zhou R, Payne ME, Bales CW. Improved Function With Enhanced Protein Intake per Meal: A Pilot Study of Weight Reduction in Frail, Obese Older Adults. J Gerontol A Biol Sci Med Sci. 2016 Oct;71(10):1369-75. doi: 10.1093/gerona/glv210. Epub 2016 Jan 18. PMID 26786203
- [Derived] McDonald SR, Porter Starr KN, Mauceri L, Orenduff M, Granville E, Ocampo C, Payne ME, Pieper CF, Bales CW. Meal-based enhancement of protein quality and quantity during weight loss in obese older adults with mobility limitations: rationale and design for the MEASUR-UP trial. Contemp Clin Trials. 2015 Jan;40:112-23. doi: 10.1016/j.cct.2014.11.010. Epub 2014 Nov 20. PMID 25461495